CLINICAL TRIAL: NCT02660619
Title: Validation of PRISM-5-Op, Measure Of Addiction To Prescription Opioid Medication
Status: Completed | Type: Observational
Sponsor: Member Companies of the Opioid PMR Consortium (Industry)
Collaborators: Research Foundation for Mental Hygiene, Inc. (Other); Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: Observational Study 3033-5; Study 3033-5 (Other: Member Companies of the Opioid PMR Consortium)
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Opioid-Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Low-risk patients: These will be patients with a prescription for opioids for chronic pain for at least 30 days, recruited from university-affiliated pain and rehabilitation medicine clinics that routinely employ precautions to avoid prescribing such medication to individuals seeking it for non-therapeutic reasons
  Interventions: Other: Psychiatric Research Interview for Substance and Mental Disorders (PRISM-5-Op)
- High-risk patients: These patients will be in treatment for addiction to opioids and have (or have had) a prescription of opioids to treat pain.
  Interventions: Other: Psychiatric Research Interview for Substance and Mental Disorders (PRISM-5-Op)

INTERVENTIONS:
Other: Psychiatric Research Interview for Substance and Mental Disorders (PRISM-5-Op)

SUMMARY:
The purpose is to validate the PRISM-5-Op as a measurement of prescription opioid substance use disorder.

DETAILED DESCRIPTION:
"Based on a review of the literature, the Food and Drug Administration (FDA) concluded that more data are needed regarding the serious risks of misuse, abuse, addiction, overdose, and death associated with the long-term use of extended release/long acting (ER/LA) opioid analgesics. Thus, the FDA is requiring that ER/LA opioid analgesic drug sponsors conduct post-marketing studies to assess these risks. The present study, PMR Study #2065-2, focuses on addiction, and addresses the FDA requirement to conduct a validation study of the measure of addiction that will be used in PMR Study #2065-1.

The primary objective for Study 2b is to validate PRISM-5-Op measures of DSM-5 prescription opioid SUD/addiction in patients who have, or have had, a prescription for opioids for at least 30 days to treat chronic pain"

ELIGIBILITY:
Inclusion Criteria:

1. Has or has had a prescription for opioids for chronic pain for at least 30 days
2. Age 18 years or older and English-speaking
3. Willing and able to provide informed consent"

Exclusion Criteria:

1. Patient has a hearing or vision impairment that would preclude an interview or completion of self-administered questionnaires
2. Patient too cognitively impaired to give informed consent or participate in the evaluations.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from low-risk and high-risk treatment settings in the greater New York City metropolitan area, which includes the five boroughs of the city and Long Island. Thus, the population will be a mix of urban and suburban participants.
Sampling Method: Non-Probability Sample
Enrollment: 606 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Diagnoses of Addiction to Prescription Opioids via PRISM-5-Op | Up to 14 days (reliability determined by re-interviews 1-14 days after first interview)
  PRISM-5-Op diagnoses of DSM-5 SUD/addiction to prescription opioids. These diagnoses will be in two forms: unadjusted, meaning that the criteria will be rated positive if present without regard to the intent of the behavior, and adjusted, i.e., that criteria will be rated positive only if structured evaluation indicates that they represent addiction indicators (non-therapeutic intent) rather than treatment of pain (therapeutic intent).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R Petronis, Study Chair — Pfizer

REFERENCES:
- [Derived] Hasin DS, Shmulewitz D, Stohl M, Greenstein E, Aharonovich E, Petronis KR, Von Korff M, Datta S, Sonty N, Ross S, Inturrisi C, Weinberger ML, Scodes J, Wall MM. Diagnosing Prescription Opioid Use Disorder in Patients Using Prescribed Opioids for Chronic Pain. Am J Psychiatry. 2022 Oct;179(10):715-725. doi: 10.1176/appi.ajp.21070721. Epub 2022 Jun 15. PMID 35702830